CLINICAL TRIAL: NCT06094491
Title: VIDA: Virtual Diabetes Group Visits Across Health Systems: Randomized Control Trial
Brief Title: Virtual Diabetes Group Visits Across Health Systems
Acronym: VIDA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Wake Forest University Health Sciences (Other); ACCESS Community Health Network (Other); Midwest Clinicians' Network (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB23-0325; P50MD017349-04 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-07

CONDITIONS: T2DM (Type 2 Diabetes Mellitus); Hypertension; Heart Disease Chronic; Stroke; Hyperlipidemias; Peripheral Vascular Diseases; Obesity
Keywords: virtual group visits
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Stroke; Hyperlipidemias; Peripheral Vascular Diseases; Obesity

STUDY DESIGN:
Intervention Model Description: Type I hybrid effectiveness-implementation cluster randomized trial among adult patients with T2DM across 9 intervention sites and 9 control sites
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Group Visit Arm (Experimental): These subjects will attend 6 monthly virtual group visits hosted by ACCESS or Advocate research staff.
  Interventions: Behavioral: Virtual Group Visit
- Usual Care Arm (No Intervention): These subjects will receive usual diabetes care at ACCESS or Advocate health centers.

INTERVENTIONS:
Behavioral: Virtual Group Visit — Group visits must have these core components: diabetes education, group social support and goal setting.
  Arms: Virtual Group Visit Arm

SUMMARY:
The purpose of this project is to evaluate the effectiveness of a virtual diabetes group visits on patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Managing diabetes can be complex and burdensome; patients must modify their diet, take medications, check their blood sugar, and visit their healthcare providers regularly. Diabetes group visits (GVs)-virtual group education and diabetes support, including goal setting-create a unique setting where patients can connect with peers and receive medical care and support. GVs can improve glycemic control and decrease healthcare utilization. GVs can provide patients with comprehensive care for their multimorbid chronic condition.

Virtual GVs provide an opportunity to adapt to the current trends of telehealth and the ability to increase reach and scalability across multiple sites. Before the model can be widely adopted, important questions about the effectiveness and implementation of the virtual diabetes GV model need to be addressed. The investigators propose to build on an established program of diabetes GVs. This proposal aims to implement the virtual GV model (VIDA: Virtual Diabetes Group Visits Across Health Systems) in two distinct health systems in the Chicago region. Access Community Health Network (ACCESS) is one of the largest federally qualified health centers (FQHCs) in the United States with 35 sites across the Chicago metropolitan area, providing care for 175,000 medically under-resourced and low-income patients each year. Advocate Health Care (ADVOCATE) is a large, integrated private not-for-profit health system that includes 26 hospitals and more than 500 ambulatory sites. The system provides care across more than 129 primary care clinics in Illinois serving over 117,000 patients. Both are community-based health systems serving low-income communities in Chicago and are network partners of the Chicago Chronic Conditions Engagement Network (C3EN).

No studies have systematically implemented virtual diabetes GVs for adults with T2DM in the real-world primary care setting or across distinct health systems. The ability to train, implement, and evaluate virtual GVs across systems with different care models provides the opportunity to learn about adaptation and the obstacles and facilitators for implementation. This proposed study will compare virtual diabetes GVs to usual care using a type I hybrid effectiveness-implementation design via a pragmatic cluster randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient at a PARTICIPATING clinic (at least one visit in year prior to first GV)
* Type 2 diabetes
* ≥ 18 years old
* A1C>8% within 6 months prior to first GV (we will first recruit patients with A1C>9%, then if spaces still available A1C>8.5%, then if spaces still available A1C>8%)
* At least one additional cardiovascular condition (hypertension, heart disease, stroke, hyperlipidemia, peripheral vascular disease, or BMI ≥ 30)
* English or Spanish speaking
* PCP assented to recruiting patient
* Patient provides written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
A1c | 12 months
  This is blood test that measures the percent of glucose and hemoglobin bound together.

SECONDARY OUTCOMES:
Systolic blood pressure | 12 months
  Systolic blood pressure measures the arterial pressure
Body Mass Index | 12 months
  Measure of body fat based on height and weight
Low density lipoproteins | 12 months
  a measure of cholesterol in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Arshiya Baig, MD, Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Access Community Health Network, Chicago, Illinois
  - Advocate Health Care, Orland Park, Illinois

IPD SHARING:
Plan to Share IPD: No